CLINICAL TRIAL: NCT05716555
Title: Safety and Efficacy of Deep Brain Stimulation for Treatment Resistant Depression
Brief Title: Deep Brain Stimulation for Treatment Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Hemmings Wu, Neurosurgeon, Assistant Professor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR2021001074
Record Dates: First submitted 2022-12-19; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Depressive Disorder, Major
Keywords: deep brain stimulation; lateral habenula
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Deep brain stimulation — Electrical stimulation of lateral habenula

SUMMARY:
This study will investigate the safety and efficacy of deep brain stimulation (DBS) in lateral habenula (LH) for patients with treatment-resistant depression.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70, regardless of gender;
2. Diagnostic And Statistical Manual Of Mental Disorders 5th Ed (DSM-V), for Psychiatrists' Examination of Severe Depressive Disorders;
3. Same diagnostic conclusions based on DSM-V made by two independent psychiatrists;
4. A minimum of 24 months of depressive history, over 2 or more adequate antidepressant trials with Hamilton Depression Rating Scale (HAMD) reduction rate ≤20% (including MECT) ;
5. HAMD-17 scores ⩾ 20 at screening;
6. Functional General Assessment Table (GAF) rating ≤50;
7. Able to comply with the operational and administrative requirements of participation in the study, and able to give written informed consent.

Exclusion Criteria:

1. Patients with severe or unstable mental, liver, kidney, endocrine, hematological diseases, or those with psychotic co-morbidities, including personality disorders;
2. History of substance abuse in the past 12 months; history of epilepsy, or febrile seizure in childhood;
3. Patients who have attempted suicide within the past 6 months, or have had a secondary suicide attempt within the past 2 years;
4. Women who are breastfeeding, pregnant, or intend to be pregnant during the clinical study;
5. Any surgical contraindications to undergoing deep brain stimulation (DBS);
6. Patients who cannot give full informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2021-03-14 (Actual); Primary Completion 2023-03-13 (Estimated); Study Completion 2024-03-13 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 52 weeks after surgery
  Change in Hamilton Depression Rating Scale score from baseline to 52 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University School of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes